CLINICAL TRIAL: NCT06405516
Title: Platelet Count and Function After Usage of Two Different Cell Saver Devices During Cardiac Surgery: a Randomized Controlled Multi-center Equivalence Trial.
Brief Title: Platelet Function After Cardiac Surgery.
Acronym: PLFICS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University Hospital, Geneva (Other); University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: BASEC 2023-D0074
Record Dates: First submitted 2024-04-29; First posted 2024-05-08 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Platelet Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients undergoing cardiac surgery using the conventional cell saver device (Active Comparator)
  Interventions: Device: Autologous blood cell salvage with in-house device
- Patients undergoing cardiac surgery using the cell saver device (Experimental)
  Interventions: Device: Autologous cell salvage with i-Sep SAME device

INTERVENTIONS:
Device: Autologous blood cell salvage with in-house device — In addition to standard procedures in this patient population, study participants will receive point-of-care analysis of platelet function and coagulation (laboratory analysis and viscoelastic tests, if not already provided by the responsible anesthesiologist) based on the clinical situation, at different time points before and after retransfusion of processed cell salvage blood.
  Arms: Patients undergoing cardiac surgery using the conventional cell saver device
Device: Autologous cell salvage with i-Sep SAME device — In addition to standard procedures in this patient population, study participants will receive point-of-care analysis of platelet function and coagulation (laboratory analysis and viscoelastic tests, if not already provided by the responsible anesthesiologist) based on the clinical situation, at different time points before and after retransfusion of processed cell salvage blood.
  Arms: Patients undergoing cardiac surgery using the cell saver device

SUMMARY:
Intraoperative cell salvage is commonly used in cardiac surgery to reduce the administration of allogeneic red blood cells and thus improve the outcome for the patient. When processing the salvaged blood, however, a large part of the patient's plasma is washed out. This is a disadvantage with regard to an optimal coagulation situation after cardiac surgery.

There are currently various cell saver systems on the market. According to the manufacturers, the plasma is returned to the patient in different quantities as part of the processing procedure. Thus, it can be assumed that in addition to red blood cells, platelets (part of plasma) are retransfused and contribute to an optimized coagulation. Unfortunately, there is a lack of studies in this regard in the cardiac surgery population.

The investigators aim to study the performance of two different cell saver devices regarding preservation of platelet number and function.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Elective high risk cardiac surgery with cardiopulmonary bypass usage
* Cardiopulmonary bypass time > 120 minutes
* Written informed consent

Exclusion Criteria:

* Preoperative use of oral or intravenous anti-coagulants or antiplatelet agents (except aspirin)
* Inability to understand and sign the informed consent form (e.g. language problems, dementia, mental disorders).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Platelet number | Perioperative period (begins on the day of surgery and ends on the day after surgery)
  Platelet number as measured by flow cytometry after processing and retransfusion of the salvaged blood to the patient.

SECONDARY OUTCOMES:
Platelet function measured by multiple electrode aggregometry | Perioperative period (begins on the day of surgery and ends on the day after surgery)
  Platelet function, as measured by point-of-care test
Platelet function measured by platelet activation markers (P-selectin) | Perioperative period (begins on the day of surgery and ends on the day after surgery)
  Platelet function, as measured by point-of-care test
Platelet function measured by platelet activation markers (GPIb and GPIIb) | Perioperative period (begins on the day of surgery and ends on the day after surgery)
  Platelet function, as measured by point-of-care test
Platelet function measured with viscoelastic point-of-care test (Clotpro) | Perioperative period (begins on the day of surgery and ends on the day after surgery)
  Platelet function, measured by point-of-care test using ExTest und FibTest assays with viscoelastic point-of-care test device
Platelet function measured with viscoelastic point-of-care test (ROTEM) | Perioperative period (begins on the day of surgery and ends on the day after surgery)
  Platelet function, measured by point-of-care test using ExTEM und FibTEM assays with viscoelastic point-of-care test device
Number of allogeneic blood products transfused | Perioperative period (begins on the day of surgery and ends on the day after surgery)
  Number of allogeneic blood products used (red blood cell, fresh frozen)

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Erdoes, MD, Study Chair — University of Bern
Locations (1):
- Department of Anesthesiology and Pain Medicine, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No